CLINICAL TRIAL: NCT06607666
Title: Acromegaly Resistant to Conventional Dose of First Generation Somatostatin Ligands
Acronym: ACRO-SSA
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 5132
Record Dates: First submitted 2023-03-06; First posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Acromegaly
MeSH Terms: conditions — Acromegaly

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Low dose to fg-SRLs: Patients responsive to low dose to fg-SRLs
  Interventions: Drug: Lanreotide autogel
- High dose to fg-SRLs: Patients responsive to high dose to fg-SRLs
  Interventions: Drug: Lanreotide autogel
- Other treatments: Patients not responsive to low/high dose of fg-SRLs
  Interventions: Drug: Lanreotide autogel

INTERVENTIONS:
Drug: Lanreotide autogel — Identification of clinical, biochemical, molecular markers of response to low and high dose of fg-SRLs
  Other Names: Somatostatin Receptor ligand

SUMMARY:
Acromegaly is a chronic disease, with a high frequency of systemic complications and reduced life span, in cases of persistently active disease. The remission of acromegaly through the surgical removal of the pituitary adenoma ranges from the 10 to 70%, according to surgery experience, tumor invasion and dimension. The medical treatment can reach the control of acromegaly disease in around 35-45% of patients treated with first generation somatostatin analogues (first gen-SSAs) at standard dose. Instead, patients partially or completely resistant to treatment with first gen-SSAs may reach the control of acromegaly by treatments with high dose/frequency first gen-SSAs, antagonist of GH receptor and second generation SSAs. At the actual moment, the scientific societies are heavily working for reaching definitive guidelines for the management of second line treatments in acromegaly patients resistant to first gen-SSAs at standard dose. According to the most recent expert opinions, consensus and guidelines, the choice of second line treatment may be oriented by patients' comorbidities and molecular characterization of the GH secreting tumors. However, a consensus of the clinical use of molecular biomarkers was not reached.

The primary objective of this study is to define the number of patients who had reached the control of acromegaly at 6, 12 and 24 months of treatment, according to the following two treatment schemes (Lanreotide ATG at conventional dose versus Lanreotide ATG at high dose/frequency). The secondary objectives are to evaluate the role of the tumor molecular biomarkers, clinical and biochemical features of acromegaly and of morphological features of GH secreting tumors in predicting the outcome of the previous detailed two treatment schemes.

For reaching these aims, we designed an observational, retrospective, mono-center study on acromegaly patients. Patients will be enrolled according to strict inclusion/exclusion criteria. Data collection will be retrospectively conducted on molecular biomarkers (e.g. genomic polymorphism of the gene of the GH receptor on patients' blood; expression of GH, prolactin, Ki-67 labeling index (Li), p53, subtype 2 and 5 of the somatostatin receptor, cytokeratin pattern and number of mitosis through immunohistochemistry on paraffin-fixed samples of the patients' pituitary GH secreting tumors) and on clinical (e.g. gender and age at acromegaly diagnosis) and biochemical features (e.g. random GH, cycle GH and GH nadir, IGF-I, prolactin values at the time of acromegaly diagnosis, after pituitary surgery and before starting treatment with first gen-SSAs). The results of these clinical, biochemical and morphological markers will be correlated to the outcome of treatment with Lanreotide ATG, both at standard dose and at high dose/high frequency.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed for acromegaly;
* patients underwent first line treatment for acromegaly with pituitary surgery;
* patients with acromegaly diagnosis confirmed through the pathological examination of the resected pituitary tumor;
* patients affected by persistently active acromegaly, after pituitary surgery and consecutively treated with Lanreotide ATG at standard dose;
* patients treated with Lanreotide ATG at standard dose for at least 12 consecutive months and/or patients treated with Lanreotide ATG at standard dose for 6 consecutive months and then at high dose/frequency for at least 12 consecutive month;
* cases with available of all data, required for this study in internal database.

Exclusion Criteria:

* patients underwent medical therapies or radiotherapy before pituitary surgery;
* patients underwent radiotherapy within 3 years before starting the treatment with Lanreotide ATG;
* patients on treatment with other drugs for acromegaly as dopamine agonist and/or antagonist of GH receptor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 150 acromegaly patients
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2023-01-26 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Lanreotide ATG efficacy | 24 months
  number of patients who had reached the control of acromegaly at 6, 12 and 24 months of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Sabrina Chiloiro, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS, UOC ENDOCRINOLOGIA, Roma, Italy